CLINICAL TRIAL: NCT04562662
Title: Evaluation of mediVR-KAGURA Guided Therapy: A Prospective Interventional Study
Brief Title: Evaluation of mediVR-KAGURA Guided Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Japan Society of Clinical Research (Other)
Responsible Party: Principal Investigator, Masahiko Hara, Principal Investigator, Japan Society of Clinical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202001
Record Dates: First submitted 2020-09-12; First posted 2020-09-24 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Physical Disability; Cognitive Dysfunction
Keywords: Virtual Reality; Physical; Cognitive
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Single arm (all participants receive interventions)
  Interventions: Device: mediVR KAGURA

INTERVENTIONS:
Device: mediVR KAGURA — Approximately 20 min mediVR KAGURA-guided rehabilitation

SUMMARY:
The objective is to evaluate mediVR-KAGURA guided therapy for the treatments of physical and cognitive dysfunctions regardless of baseline disease in a prospective interventional design.

DETAILED DESCRIPTION:
The patients sit on an upright chair, wear a head-mounted display (HMD) and grab two handheld controllers in a motion-tracked three-dimensional space called "room scale" of the mediVR-KAGURA (mediVR, Inc. Toyonaka City, Osaka, Japan). mediVR-KAGURA can provide users with >90 frames per second (fps) graphic operation with an approximately 110° viewing angle and accurate three-dimensional tracking technology.

First, we evaluate conventional and maximum reaching distances at 0°, 45°, and 90° level surface for the left hand (0L, 45L, 90L) and at 90°, 135°, and 180° level surface for the right hand (90R, 135R, or 180R) for calibration in a sitting position. During rehabilitation, patients are instructed to touch a fixed objects or catch a falling objects at the pre-specified height and distance levels in each degree. Horizontal distances were classified into three categories, namely long, middle, and short which were calculated using the following formulas: 0.9 * maximum reaching distance, 0.9 * (conventional + maximum reaching distances)/2, and conventional reaching distance respectively. A falling object disappeared at a 20 cm height for safety if the patients missed to catch it. The purpose of reaching hands was to stimulate and break down body trunk balance, and to train participants to balance for stable walking. By thinking about the timing and distance and recognizing the next targets repeatedly, cognitive function was simultaneously stimulated for dual-task training.

The 7 parameters of the rehabilitation programs can be set like as follows: (1) distance (short, middle or long), (2) direction (0L, 45L, 90L, 90R, 135R, or 180R), (3) height of object, (4) size of object (center or outline), (5) size of sensing sphere of the controller, (6) falling speed of the square box (from 0 to 300 cm/s), and (7) intervals for each task. Participants first underwent practical programs to familiarize themselves with mediVR-KAGURA guided rehabilitation, followed by rehabilitation programs. Provision of the rehabilitation programs will be personalized.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with physical and/or cognitive dysfunctions
2. Agreed to the participation of this study with written informed consent by themselves or guardians

Exclusion Criteria:

1. Inappropriate candidates at attending physician's discretion

Ages: 6 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Timed up and go test | baseline (pre-intervention), immediately after the first intervention, average of 1, 3 and 6 months after the intervention
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. Shorter score means a better outcome. The minimum value could be 5 seconds or less, and the maximum value could be infinity (cannot complete the test).
Change in Trail Making Test | baseline (pre-intervention), immediately after the first intervention, average of 1, 3 and 6 months after the intervention
  The Trail Making Test (TMT) is a neuropsychological test of visual attention and task switching. Shorter score means a better outcome. The minimum value could be 15 seconds or less, and the maximum value could be infinity or be defined as 300 seconds when patients cannot complete the test.

SECONDARY OUTCOMES:
Changes in Functional Independence Measure | baseline (pre-intervention), immediately after the first intervention, average of 1, 3 and 6 months after the intervention
  The Functional Independence Measure (FIM) is an assessment tool that aims to evaluate the functional status of patients throughout the rehabilitation process following a stroke, traumatic brain injury, spinal cord injury or cancer. Higher score means a better outcome. The minimum value is 18, and the maximum value is 126.
Changes in Berg balance scale | baseline (pre-intervention), immediately after the first intervention, average of 1, 3 and 6 months after the intervention
  The Berg Balance Scale (or BBS) is a widely used clinical test of a person's static and dynamic balance abilities. Higher score means a better outcome. The minimum value is 0, and the maximum value is 56.
Changes in Mini Mental State Examination | baseline (pre-intervention), immediately after the first intervention, average of 1, 3 and 6 months after the intervention
  The Mini-Mental State Examination (MMSE) test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Higher score means a better outcome. The minimum value is 0, and the maximum value is 30.
Changes in Self Rating Depression Scale | baseline (pre-intervention), immediately after the first intervention, average of 1, 3 and 6 months after the intervention
  The Self Rating Depression Scale (SDS) is a psychiatric measuring instrument having descriptive words and phrases that indicate the severity of depression for a time period. Lower score means a better outcome. The minimum value is 20, and the maximum value is 80.

CONTACTS AND LOCATIONS:
Overall Officials: Masahiko Hara, MD, PhD, Study Chair — Cloud Clinic
Locations (1):
- Cloud Clinic, Takarazuka, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No